CLINICAL TRIAL: NCT02081495
Title: A Pivotal Bioequivalence Study of DOXIL®/CAELYX® Manufactured at a New Site in Subjects With Advanced or Refractory Solid Malignancies Including Subjects With Ovarian Cancer
Brief Title: A Study of DOXIL/CAELYX in Patients With Advanced or Refractory Solid Malignancies Including Patients With Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR103500; DOXILNAP1004 (Other: Janssen Research & Development, LLC); 2013-004641-16 (EudraCT Number)
Record Dates: First submitted 2014-03-05; First posted 2014-03-07 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-10

CONDITIONS: Neoplasms
Keywords: Neoplasms; Neoplasms, Ovarian; Ovarian Cancer; Advanced or Refractory Solid Malignancies; Doxorubicin; DOXIL; CAELYX
MeSH Terms: conditions — Neoplasms; Ovarian Neoplasms | interventions — liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence AB (Experimental): Twenty-one participants will receive DOXIL/CAELYX reference product in Cycle 1 and DOXIL/CAELYX test product in Cycle 2. Each cycle will be separated by 28 days.
  Interventions: Drug: DOXIL/CAELYX reference product (Treatment A); Drug: DOXIL/CAELYX test product (Treatment B)
- Sequence BA (Experimental): Twenty-one participants will receive DOXIL/CAELYX test product in Cycle 1 and DOXIL/CAELYX reference product in Cycle 2. Each cycle will be separated by 28 days.
  Interventions: Drug: DOXIL/CAELYX reference product (Treatment A); Drug: DOXIL/CAELYX test product (Treatment B)

INTERVENTIONS:
Drug: DOXIL/CAELYX reference product (Treatment A) — Participants will receive DOXIL/CAELYX reference product 50 mg/m2 as an intravenous (into a vein) infusion over 90 minutes on Day 1.
  Other Names: DOXIL; CAELYX
Drug: DOXIL/CAELYX test product (Treatment B) — Participants will receive DOXIL/CAELYX test product 50 mg/m2 as an intravenous infusion over 90 minutes on Day 1.
  Other Names: DOXIL; CAELYX

SUMMARY:
The purpose of this study is to support the qualification of a replacement manufacturing site for DOXIL/CAELYX.

DETAILED DESCRIPTION:
This is a randomized (study medication is assigned by chance), open-label (all people know the identity of the intervention), single dose, 2-cycle, crossover (method used to switch participants from one treatment arm to another in a clinical study), and bioequivalence (biological equivalence of two formulations of a study medication) study of DOXIL/CAELYX in participants with advanced or refractory solid malignancies (including at least 24 participants with ovarian cancer). This study has an adaptive 2-stage design. Bioequivalence based on encapsulated doxorubicin will be tested at the end of Stage 1 using data from at least 24 participants with ovarian cancer. An interim analysis of free doxorubicin will be performed at the end of Stage 1 using data from 42 participants of all cancer types. The study may continue into Stage 2 with additional participants of all cancer types; and final evaluation of bioequivalence for free doxorubicin will be performed at the end of Stage 2. The study will include a screening phase (within 28 days before the first study medication administration) followed by the treatment phase consisting of 2 doxorubicin treatment cycles (28 days each) and an end-of-treatment visit on Day 58. Participants may enter an optional extension phase after 2 cycles. Safety will be evaluated by the assessment of adverse events, vital signs, 12-lead electrocardiogram, clinical laboratory testing, and left ventricular ejection fraction (measurement of the percentage of blood leaving the heart each time when it contracts) throughout the study. Blood samples for pharmacokinetic analysis will be obtained from all participants at specified times over 29 days after starting each study drug administration in Cycles 1 and 2 for determination of plasma concentrations of encapsulated and free doxorubicin.

ELIGIBILITY:
Inclusion Criteria:

* Having advanced or refractory solid malignancies (histologically or cytologically confirmed advanced ovarian cancer failing platinum-based chemotherapy or metastatic breast cancer after failing approved life prolonging therapies or any solid malignancy that is metastatic or unresectable, and for which standard treatment is no longer an option)
* Eastern cooperative oncology group performance status 0 to 2
* Recovered from the acute toxicity (except alopecia and asymptomatic neuropathy) of any prior treatment
* Participants with prior doxorubicin (or other anthracyclines) or without any prior anthracylin exposure can also be included
* Agrees to protocol-defined use of effective contraception

Exclusion Criteria:

* Positive history of known brain metastases or leptomeningeal disease (spreading of cancer throughout the protective membranes covering the brain and spinal cord). Participants with brain metastases can only be enrolled if the following conditions are all met: 1) Brain metastases have been treated and stable for more than 4 weeks, 2) No evidence for progression or hemorrhage after treatment, 3) Steroid treatment was discontinued at least 2 weeks prior to first administration of DOXIL/CAELYX, and 4) Enzyme inducing anti-epileptic medicines were discontinued at least 4 weeks before first administration of DOXIL/CAELYX
* Use of an investigational medicine within 21 days or 5 half-lives (whichever is shorter) prior to the first dose of DOXIL/CAELYX
* Any major surgery, radiotherapy, or immunotherapy within the last 21 days. Chemotherapy regimens with delayed toxicity within the last 3 weeks (or within the last 6 weeks for prior nitrosourea or mitomycin C)
* Unstable angina or myocardial infarction within the preceding 12 months; congestive heart failure or any history of uncontrolled cardiac disease
* Having an uncontrolled infection and uncontrolled concurrent illness including, but not limited to, poorly controlled hypertension or diabetes, or psychiatric illness/social situation that may potentially impair the participant's compliance with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of encapsulated doxorubicin | Predose, and postdose Day 1 (Minutes 15, 30, 60, 90, 95, 105; Hours 2, 3, 4, 6, 8), Days 2, 3, 4, 5, 8, 15, 22, and 26 (for Cycles 1 and 2)
  Cmax is defined as the maximum observed analyte concentration.
Time to reach the maximum observed plasma concentration (Tmax) of encapsulated doxorubicin | Predose, and postdose Day 1 (Minutes 15, 30, 60, 90, 95, 105; Hours 2, 3, 4, 6, 8), Days 2, 3, 4, 5, 8, 15, 22, and 26 (for Cycles 1 and 2)
  Tmax is defined as the actual sampling time to reach maximum observed analyte concentration.
Area under the plasma concentration-time curve from time 0 to infinite time (AUC[0-infinity]) of encapsulated doxorubicin | Predose, and postdose Day 1 (Minutes 15, 30, 60, 90, 95, 105; Hours 2, 3, 4, 6, 8), Days 2, 3, 4, 5, 8, 15, 22, and 26 (for Cycles 1 and 2)
  AUC(0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of the Area Under the Curve (AUC) last and AUC(last)/lambda, in which AUC(last) is the last observed quantifiable concentration.

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of free doxorubicin | Predose, and postdose Day 1 (Minutes 15, 30, 60, 90, 95, 105; Hours 2, 3, 4, 6, 8), Days 2, 3, 4, 5, 8, 15, 22, and 26 (for Cycles 1 and 2)
  Cmax is defined as maximum observed analyte concentration.
Time to reach the maximum observed plasma concentration (T max) of free doxorubicin | Predose, and postdose Day 1 (Minutes 15, 30, 60, 90, 95, 105; Hours 2, 3, 4, 6, 8), Days 2, 3, 4, 5, 8, 15, 22, and 26 (for Cycles 1 and 2)
  Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Area under the plasma concentration-time curve from time 0 to infinite time (AUC[0 - infinity]) of free doxorubicin | Predose, and postdose Day 1 (Minutes 15, 30, 60, 90, 95, 105; Hours 2, 3, 4, 6, 8), Days 2, 3, 4, 5, 8, 15, 22, and 26 (for Cycles 1 and 2)
  AUC(0-infinity) is area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of Area under Curve (AUC) last and AUC(last)/lambda, in which AUC(last) is the last observed quantifiable concentration.
Number of participants with adverse events as a measure of safety and tolerability | Up to Day 86
Number of participants with response to the study medication at End-of-Treatment visit (Day 58) | Day 58 or 30 days after the last dose of the study medication for early withdrawal participants
  The investigator will determine the response to the study medication as Complete Response (CR), Partial Response (PR) or Stable Disease (SD) according to the Response Evaluation Criteria in Solid Tumors (RECIST). As per the RECIST, CR is defined as the disappearance of all target and non-target lesions, PR is defined as 30% or more decrease in the sum of longest diameter of all target lesions from the baseline sum; and SD is defined as none of the CR and PR.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (6):
- Los Angeles, California, United States
- Belgium (2):
  - Brussels
  - Wilrijk
- Edmonton, Alberta, Canada
- Spain (2):
  - Barcelona
  - Madrid

REFERENCES:
- See also: A Pivotal Bioequivalence Study of DOXIL®/CAELYX® Manufactured at a New Site in Subjects with Advanced or Refractory Solid Malignancies — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=6195&filename=CR103500_CSR.pdf